CLINICAL TRIAL: NCT04960540
Title: Multimodal Brain Imaging Study of Language Cognitive Function in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Multimodal Brain Imaging Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018273
Record Dates: First submitted 2021-06-27; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- impaired speech comprehension processing in ALS: Brain functional network mechanism of impaired speech comprehension processing in ALS
  Interventions: Other: MRI,
- language use processing injury in ALS: Brain functional network mechanism of language use processing injury in ALS
  Interventions: Other: MRI,
- motor executive processing injury in ALS: Brain functional network mechanism of motor executive processing injury in ALS
  Interventions: Other: MRI,
- anguage cognitive impairment in ALS: Brain structural network mechanism of language cognitive impairment in ALS
  Interventions: Other: MRI,

INTERVENTIONS:
Other: MRI, — In this project, multi-modal brain imaging methods, such as resting-state functional MRI, task-state functional MRI, structural MRI and diffusion tensor imaging, will be used to analyze brain structure, gray matter morphology, white matter fibrous brain functional activation mode and brain functional connectivity network, and other dimensions.
  In particular, combined with the brain functional activities of ALS patients in the cognitive processing task of language understanding and language use, the brain network damage of ALS patients in motor and executive function was compared, and the neural activities and network mechanism of specific changes in language cognitive processing in ALS patients were investigated. Combined with the clinical neuropsychological behavior evaluation data

SUMMARY:
To explain the key brain network nodes and their brain mechanisms of ALS language cognitive impairment and decline, reveal the neural mechanism of the association between ALS language cognitive impairment and motor executive function, and provide potential early diagnostic markers and targeted therapeutic targets for ALS language cognitive impairment.

DETAILED DESCRIPTION:
【 Objective 】 To elucide the key brain network nodes and their brain mechanisms of language cognitive impairment and decline in ALS, and to reveal the neural mechanism of the association between language cognitive impairment and motor executive function in ALS, so as to provide potential early diagnostic markers and targeted therapeutic targets for language cognitive impairment in ALS.

[Design] With the help of multi-modal brain imaging methods such as resting-state functional MRI, task-state functional MRI, structural MRI and diffusion tensor imaging, this project will analyze from multiple dimensions such as brain structure, gray matter morphology, white matter fibrous brain functional activation mode and brain functional connectivity network.

In particular, combined with the brain functional activities of ALS patients in the cognitive processing task of language understanding and language use, the brain network damage of ALS patients in motor and executive function was compared, and the neural activities and network mechanism of specific changes in language cognitive processing in ALS patients were investigated. Combined with the clinical neuropsychological behavior evaluation data, To deeply understand the neural mechanism of language cognitive impairment in ALS patients.

The research will be divided into four parts, including: the brain functional network mechanism of ALS language understanding processing injury, ALS language use processing injury, ALS motor executive processing injury, ALS language cognitive injury brain structural network mechanism.

Ten patients with ALS were included in each part of the study, and 40 patients with ALS in four parts were included in the study. Multimodal magnetic resonance scanning and cognitive assessment were performed.

Normal healthy controls for this study will be provided by the research team of Peking University Magnetic Resonance Imaging Research Center of this project group.

ELIGIBILITY:
Inclusion Criteria:

* Entry criteria:

  1. Satisfied clinically possible ALS, laboratory supported suspected ALS, clinically suspected ALS or clinically confirmed ALS in the diagnostic criteria of ALS EL Escorial revised in 1998
  2. Ages 18-70
  3. Agree and sign the informed consent

Exclusion Criteria:

* 1) Severe respiratory dysfunction, unable to cooperate with NMR examination 2) Severe dysarthria and limb dysfunction, unable to cooperate with the neuropsychological examination 3) Patients with absolute or relative contraindications to MRI, including: a) Patients with cardiac pacemakers, cochlear implants, built-in pumps, nerve stimulators, artificial metal heart valves, etc.; B) After ligation of aneurysm clip (except non-paramagnetic, such as titanium alloy); C) Internal ferromagnetic metal implants (excluding metal IUD and fixed dentures); D) Claustrophobic; E) Patients with epilepsy 4) Pregnant patients 5) illiterate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (I) Study population
  1. Inclusion criteria:
  1. Satisfied clinically possible ALS, laboratory supported suspected ALS, clinically suspected ALS or clinically confirmed ALS in the diagnostic criteria of ALS EL Escorial revised in 1998
  2. Ages 18-70
  3. Agree and sign the informed consent
  2. Exclusion criteria:
  1. Severe respiratory dysfunction, unable to cooperate with NMR examination
  2. Severe dysarthria and limb dysfunction, unable to cooperate with the neuropsychological examination
  3. Patients with absolute or relative contraindications to MRI, including: a) Patients with cardiac pacemakers, cochlear implants, built-in pumps, nerve stimulators, artificial metal heart valves, etc.; B) After ligation of aneurysm clip (except non-paramagnetic, such as titanium alloy); C) Internal ferromagnetic metal implants (excluding metal IUD and fixed dentures); D) Claustrophobic; E) Patients with epilepsy
  4. Pregnant patients
  5. illiterate
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
ALSFRS-R score | After 1 year of recruitment
  Amyotrophic lateral sclerosis rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Shan Ye, Study Chair — Peking Yniversity Third Hospital Medical
Locations (1):
- Peking Yniversity Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No